CLINICAL TRIAL: NCT02557971
Title: Urinary Retention Rates in Clinical Practice After Treatment With OnabotulinumtoxinA for Idiopathic Overactive Bladder
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-US-OAB-0403
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BOTOX®: Patients with idiopathic overactive bladder (OAB) treated with onabotulinumtoxinA (BOTOX®) injections into the bladder as standard of care in clinical practice. No intervention was administered in this study.
  Interventions: Drug: onabotulinumtoxinA

INTERVENTIONS:
Drug: onabotulinumtoxinA — OnabotulinumtoxinA (BOTOX®) as prescribed in clinical practice.
  Other Names: BOTOX®; botulinum toxin Type A

SUMMARY:
This study is a retrospective chart review of patients treated with BOTOX® for idiopathic Overactive Bladder (OAB) as standard of care in clinical practice. The study will determine the rate of post procedural urinary retention requiring catheterization and identify factors that may predict urinary retention.

ELIGIBILITY:
Inclusion Criteria:

-Patients treated with BOTOX® for Overactive Bladder.

Exclusion Criteria:

* Received botulinum toxin formulations other than BOTOX® in the bladder.
* Had symptoms of OAB associated with a neurological condition.
* Had a history of chronic urinary retention treated with Clean Intermittent Catheterization (CIC) or indwelling catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prescribed BOTOX® for the treatment of idiopathic OAB in clinical practice.
Sampling Method: Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Post-Procedure Urinary Retention requiring Catheterization | 12 Weeks
Length of Time of Clean Intermittent Catheterization (CIC) Use | 12 Weeks

SECONDARY OUTCOMES:
Percentage of Participants with Urinary Tract Infection (UTI) | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (7):
- United States (7):
  - University of California, Davis, Davis, California
  - Capital Region Urology, Irvine, California
  - The Charlotte-Mecklenburg Hospital Authority DBA Carolinas Healthcare System, Charlotte, North Carolina
  - Alliance Urology Specialists, PA, Greensboro, North Carolina
  - Forsyth Memorial Hospital Inc. dba Novant Health Urology Partners, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Virginia Women's Center Inc., Richmond, Virginia